CLINICAL TRIAL: NCT04265222
Title: Prospective Randomized Controlled Study Utilizing the Stryker Hip-Check Software Platform
Brief Title: Cam Decompression Utilizing the Stryker Hip-Check Software Platform
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American Hip Institute (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHI-002
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Femoroacetabular Impingement
Keywords: Orthopedics; Cam Decompression; Femoroplasty; Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional Fluoroscopy (Other): Participants undergoing femoroplasty with conventional treatment
  Interventions: Other: Conventional Fluoroscopy
- HipCheck (Experimental): Participants undergoing femoroplasty with Stryker HipCheck System
  Interventions: Device: Hipcheck Software

INTERVENTIONS:
Device: Hipcheck Software — Software
  Other Names: Stryker HipCheck system
  Arms: HipCheck
Other: Conventional Fluoroscopy — Conventional Fluoroscopy
  Arms: Conventional Fluoroscopy

SUMMARY:
Accurate femoroplasty has been shown to be critical in achieving success following treatment of femoroacetabular impingement (Matsuda, Schnieder, and Sehgal 2014; Mansor et al. 2018; Larson et al. 2014). Nearly 75% of cases undergoing revision hip arthroscopy do so due to residual femoroacetabular impingement (Ricciardi et al. 2014). Femoroplasty remains one of the most challenging and time-consuming procedures in hip arthroscopy and methods to improve accuracy and optimize time management are essential. The HipCheck system is a navigational tool based on intraoperative fluoroscopy that aims at improving accuracy and efficiency of femoroplasty.

The objective of this study is to two-fold. (1) To prospectively compare surgical and (2) radiographic outcomes of patients undergoing femoroplasty with guidance of Stryker's HipCheck system to patients undergoing femoroplasty with conventional fluoroscopic methods.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively compare surgical and radiographic outcomes of patients undergoing femoroplasty with guidance of Stryker's HipCheck system to patients undergoing femoroplasty with conventional fluoroscopic methods.

Endpoints:

Time from initiation to completion of femoroplasty Accuracy of femoroplasty as determined by: alpha angle on Dunn view and AP view, femoral head offset, and area of over resection and under resection Fluoroscopic exposure (microgray and seconds) Post-operative opioid consumption/medication use

Basic design: Randomized Controlled Study

Participants: 40 patients 20 patients will undergo femoroplasty with the conventional technique 20 patients will undergo femoroplasty with the HipCheck system

Accurate femoroplasty has been shown to be critical in achieving success following treatment of femoroacetabular impingement (FAI).1-3 Nearly 75% of cases undergoing revision hip arthroscopy do so due to residual FAI. Matsuda et al. coined the term "critical corner" to describe residual impingement not resected during routine anterolateral femoroplasty. These residual cam lesions have been shown to lead to inferior outcomes and are commonly implicated in revision hip arthroscopies. These studies and others contributed to the development of the "spherical femoroplasty" as an attempt to minimize residual cam lesions while simultaneously, avoiding over-resection. Femoroplasty remains one of the most challenging and time-consuming procedures in hip arthroscopy and methods to improve accuracy and optimize time management are essential.

General Schema of Study Design Overview Patients will be randomly assigned to undergo femoroplasty either with a conventional technique or a navigational method involving the HipCheck system. Preoperatively, the patient will undergo a series of standard radiographs to assess the degree of deformity. At this time, ROM will also be assessed. During surgery time required for femoroplasty as well as total fluoroscopic exposure time, as well as total exposure in microgray will be recorded. At 2 weeks postoperatively patient will undergo a series of standard radiographs to assess accuracy of femoroplasty. Narcotic medication use, pain levels and patient-reported outcome scores (PROs) will be assessed at 2 weeks, 3 months, 6 months, and 12 months postoperatively. A clinical exam will be performed postoperatively at each visit, consisting of hip range of motion (internal/external rotation, flexion, abduction, and adduction) with the patient in the supine position, impingement tests, and gait. Radiographic measurements will be performed using the institutional PACS system as well as ImageJ for surface area calculations. The patients as well as the clinician performing postoperative radiographic calculations will be blinded to method of treatment.

The total duration of the study is 1 year and 6 months:

Legal contract & IRB review: 8 weeks Patients recruitment/procedure: 8 weeks Follow up period: 1 year Manuscript writing/submission: 8 weeks

Data Sources Research resources: Research data will be collected and recorded by study personnel designated by the Investigator.

Study Procedures

Pre-Operative A series of standard radiographs (Dunn, AP, False profile views) will be taken to understand the severity of the cam-type impingement. A clinical exam including but not limited to the following will be performed: gait (antalgic, Trendelenburg) hip range of motion (internal/external rotation, flexion, abduction, and adduction) with the patient in the supine position; anterior, posterior and lateral impingement tests; painful internal/external snapping test, FABER's test, Modified Resisted Internal rotation test, Ligamentum Teres test.

Pre-operative patient-reported outcome scores (PROs) and Visual Analog Pain Scale (VAS) will be taken during screening. The PROs include: mHHS, modified Harris Hip Score; NAHS, Nonarthritic Hip Score; iHOT-12, International Hip Outcome Tool; SF-12M, Short Form 12 Mental; SF-12P, Short Form 12-Physical; VR-12M, Veterans RAND 12-Item Health Survey Mental; VR-12P, Veterans RAND 12-Item Health Survey Physical; and Patient satisfaction (out of 10).

Intra-Operative During surgery - time required for femoroplasty as well as total fluoroscopic exposure time, as well as total exposure in microgray will be recorded. Procedural start (at initiation of femoroplasty) and finish (at completion of femoroplasty) time will be recorded for comparative analysis of both groups. Fluoroscopic exposure time and total exposure in microgray will be determined based on total number of shots taken and known duration/microgray exposure of each fluoroscopic shot. Fluoroscopic shot duration/Microgray exposure: mean total fluoroscopy time will be limited to 1.10 minutes or less (52 mGy or less per patient), based on recommendations by Budd et al. 2012

Intraoperative Fluoroscopic Image Acquisition Each patient will be placed in a neutral position to allow for the standardization and comparison with the well-centered, preoperative anteroposterior (AP) pelvic radiographs that are typically used for structural analysis and treatment planning.

Once the fluoroscopic image most closely replicates the AP pelvis, the femoral head-neck junction (FHNJ) will be assessed with fluoroscopy, with the leg in 6 different positions and fluoroscopic C-arm in 3 different positions (see table below) that allow for the evaluation of the medial and lateral FHNJ (extension views) and anterior and posterior FHNJ (flexion views). These views will be obtained by rotating the operative distal femur, flexing/extending the operative hip, and/or adducting the operative hip.

For all six positions, the angle of rotation will be verified with a Goniometer (Prestige Medical, Northridge, CA).

Measurements of the alpha angle will be performed by a single reader on each exported fluoroscopic view (corresponding to the six positions) for every control specimen with the use of the HipCheck System. For the control group the surgeon will review the fluoroscopic images prior to the resection procedure, but without making or reviewing any measurements or analysis (The HipCheck analysis platform will have "alpha angle overlay" turned off, to keep measurements from being displayed). For the HipCheck group the surgeon will review the fluoroscopic images including the HipCheck analysis for each view prior to resection.

Hip Arthroscopy (femoroplasty):

Femoroplasty will be performed using a 5.5 mm bur. This will be done in combination with the aid of fluoroscopic visualization and HipCheck technology or isolated fluoroscopic visualization, depending on the patient group assignment.

The HipCheck system will be used intraoperatively to assist with clinical decision making by assessing and providing feedback on alpha angle and confirming complete bony resection and absence of residual deformity for the test group only. To prevent over- or under resection, HipCheck provides a resection line (spline) for the surgeon to visualize and resect the desired amount, with a target alpha angle of 40 degrees.

The control group will not receive intra-operative assistance from the HipCheck software platform. Both arthroscopic and fluoroscopic imaging will be used to identify the cam and aid in resection per the standard hip arthroscopy technique.

"Postoperative" Fluoroscopic Image Acquisition At the conclusion of the hip arthroscopy, postoperative fluoroscopy views will be obtained with the same six leg positions. The angle of rotation will be verified with a Goniometer (Prestige Medical, Northridge, CA). The HipCheck tablet and software may be used to capture and later analyze the alpha angle for each of these leg positions for both the control and test groups.

Post-Operative At 2 weeks postoperatively patients will undergo a series of standard radiographs (Dunn, AP, False profile views) to assess accuracy of femoroplasty. Measurements will be performed using the institutional PACS system as well as ImageJ for surface area calculations. Accuracy of femoroplasty will be determined by: alpha angle on Dunn, AP views and false profile, femoral head offset, and area of over resection and under resection on AP. The patients as well as the clinician performing postoperative radiographic calculations will be blinded to method of treatment. A post-operative PROs and VAS Pain Score will be taken at 2 weeks, 3 months, 6 months, and 12 months post-operatively. Medication use will be documented in post-op recovery, at 2 weeks, 3months, and 12 months post-operatively. A clinical exam including range of motion assessment will be performed at 2-week, 3-, 6-, and 12-month follow-up visits.

Subject Inclusion Criteria

Candidates for this study must meet ALL of the following criteria:

1. Patients undergoing hip arthroscopy; aged 18-50 years old.
2. Radiographic evidence of a cam lesion as defined by an alpha angle greater than 60 degrees as measured on the Dunn X-ray.
3. Failure of non-conservative management

Subject Exclusion Criteria

Candidates will be excluded from the study if ANY of the following apply:

1. Unwilling to participate
2. History of prior hip conditions such as slipped capital femoral epiphysis, Legg-Calvé-Perthes disease, idiopathic avascular necrosis, hip joint trauma, and prior hip surgeries
3. The presence of a concurrent systemic inflammatory arthritis such as rheumatoid arthritis; psoriatic arthritis, ankylosing spondylitis, juvenile idiopathic arthritis, or systemic lupus erythematosus
4. Marked osteoarthritis (Tönnis grade 2 or higher)
5. Subject is considered a part of a vulnerable population
6. Pregnancy in order to avoid: x-rays and the contraindication of lying supine after 20 weeks secondary to pressure on the abdominal aorta

Subject Withdrawal Criteria Subjects may voluntarily withdraw from the study at any time for any reason. The Investigator may elect at any time to withdraw a subject from the study for any reason if such a decision is in the subject's best medical interest. If a patient discontinues the study or is withdrawn by the Investigator prior to surgery, the patient will not be counted as a completed subject and an additional subject may be enrolled to achieve the enrollment goal of 40 completed subjects.

Data Management Use established data registry and collection methodology. All preoperative and demographic data is collected and inputted into registry preoperatively. Intraoperative data and measurements are collected and inputted at time of surgery. Postoperative radiographic measurements to assess alpha angle and combined femoral offset are made within 3 months postoperatively, using a 2nd independent reader to verify inter- and intra-observer reliability.

Intraoperative data and postoperative complications are collected using OBERD system.

Risks Generalized risks to surgical procedures are present, which include but are not limited to bleeding, infection, injury to surrounding structures such as blood vessels, nerves, tendons, and bone. In addition, risks specific to hip arthroscopy include those related to hip traction related issues such as numbness and parasthesias to the perineum or soft tissue compression related complications. Lastly, risk to radiation exposure is present, however, it is limited with the use of HipCheck, as continuous fluoroscopy is not needed.

Benefits Enhanced verification of intraoperative cam resection via minimal fluoroscopic exposure. In addition, increased accuracy of cam resection with the goals of avoiding over or underresection, will thereby potentially improve patient outcomes following hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet ALL of the following criteria:

* Patients undergoing hip arthroscopy; aged 18-50 years old
* Radiographic evidence of a cam lesion as defined by an alpha angle greater than 60 degrees as measured on the Dunn X-ray.
* Failure of non-conservative management

Exclusion Criteria:

Candidates will be excluded from the study if ANY of the following apply:

* Unwilling to participate
* History of prior hip conditions such as slipped capital femoral epiphysis, Legg-Calve-Perthes disease, idiopathic avascular necrosis, hip joint trauma, and prior hip surgeries
* The presence of a concurrent systemic inflammatory arthritis such as rheumatoid arthritis; psoriatic arthritis, ankylosing spondylitis, juvenile idiopathic arthritis, or systemic lupus erythematosus
* Marked osteoarthritis (Tönnis grade 2 or higher)
* Subject is considered a part of a vulnerable population
* Pregnancy in order to avoid: x-rays and the contraindication of lying supine after 20 weeks secondary to pressure on the abdominal aorta

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
modified Harris Hip Score | 1 year
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
Nonarthritic Hip Score | 1 year
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
International Hip Outcome Tool-12 | 1 year
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
Short Form 12 Mental | 1 year
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal mental outcome
Short Form 12 Physical | 1 year
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
Veterans RAND 12-Item Health Survey Mental | 1 year
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal mental outcome
Veterans RAND 12-Item Health Survey Physical | 1 year
  Patient-reported outcome measure. Scale 0-100, 100 indicating optimal function outcome
Patient satisfaction | 1 year
  Patient-reported outcome measure. Scale 0-10, 10 indicating patient is extremely satisfied with surgery and met expectations.
Visual Analog Pain Scale | 1 year
  Patient-reported outcome measure. Scale 0-10, with 0 indicated no pain post-surgery.

SECONDARY OUTCOMES:
Age | before surgery
  Demographic information
Body Mass Index, kg/m^2 | before surgery
  Demographic information

CONTACTS AND LOCATIONS:
Overall Officials: Ajay C Lall, MD, MS, Principal Investigator — American Hip Institute
Locations (1):
- American Hip Institute, Des Plaines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larson CM, Giveans MR, Samuelson KM, Stone RM, Bedi A. Arthroscopic Hip Revision Surgery for Residual Femoroacetabular Impingement (FAI): Surgical Outcomes Compared With a Matched Cohort After Primary Arthroscopic FAI Correction. Am J Sports Med. 2014 Aug;42(8):1785-90. doi: 10.1177/0363546514534181. Epub 2014 May 29. PMID 24875469
- [Background] Mansor Y, Perets I, Close MR, Mu BH, Domb BG. In Search of the Spherical Femoroplasty: Cam Overresection Leads to Inferior Functional Scores Before and After Revision Hip Arthroscopic Surgery. Am J Sports Med. 2018 Jul;46(9):2061-2071. doi: 10.1177/0363546518779064. Epub 2018 Jun 20. PMID 29924630
- [Background] Matsuda DK, Schnieder CP, Sehgal B. The critical corner of cam femoroacetabular impingement: clinical support of an emerging concept. Arthroscopy. 2014 May;30(5):575-80. doi: 10.1016/j.arthro.2014.01.009. Epub 2014 Mar 12. PMID 24630123
- [Background] Ross JR, Larson CM, Adeoye O, Kelly BT, Bedi A. Residual deformity is the most common reason for revision hip arthroscopy: a three-dimensional CT study. Clin Orthop Relat Res. 2015 Apr;473(4):1388-95. doi: 10.1007/s11999-014-4069-9. PMID 25475714